CLINICAL TRIAL: NCT01038999
Title: Accelerated Aging, HIV Infection, Antiretroviral Therapies
Acronym: EP 45
Status: Completed | Type: Observational
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Responsible Party: Lucie Marchand/Project manager, French National Agency for Research on AIDS and Viral Hepatitis
Organization: ANRS, Emerging Infectious Diseases (Other Government)
Other Study IDs: 2008-A00905-50
Record Dates: First submitted 2009-12-23; First posted 2009-12-24 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-12

CONDITIONS: HIV Infection; Aging Accelerated; Antiretroviral Therapies
Keywords: Complementary Therapies
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- A HIV1-infected naive patients
  Interventions: Biological: Peripheral blood biological tests
- B HIV1-infected patients: in 1st line of ARV therapy for at least 12 months
  Interventions: Biological: Peripheral blood biological tests
- C= control Non infected HIV volunters
  Interventions: Biological: Peripheral blood biological tests

INTERVENTIONS:
Biological: Peripheral blood biological tests — A group and B group will be evaluated three times, at baseline, then every 12 months during 3 years. In case of initiation or changing of antiretroviral therapy, patients will be evaluated once more. Control subjects will be only evaluated at baseline.

SUMMARY:
The main goal is to confirm, among HIV1-infected patients, data from in vitro studies showing that antiretroviral therapies induce an accelerated aging through the same mechanisms than genetic laminopathies or than "physiological " aging, that is through the synthesis and persistence of farnesylated prelamin A. The secondary goal is to measure the impact of HIV infection and of antiretroviral therapies on markers of cell ageing (proteasome, mitochondria, telomere). The perspective is to fix antiretroviral therapy side effects using the same drug combination that will be used in few weeks in Marseille to treat children suffering from progeria

DETAILED DESCRIPTION:
Protease inhibitors block viral protease, as well as various other cell enzymes : ZMPSTE24 cliping off prelamin A into mature lamin A ; at least one of the Golgi proteases involved in the release of SREBP, controlling the transcription of lipid metabolism regulating genes ; mitochondrial proteases involved in the importation and further maturation of nuclear genome encoded proteins ; proteasome regulating the transcription of several genes through NF-B ; P450 cytochromes. Nucleosides inhibitors of the viral reverse transcriptase exhibit nuclear and mitochondrial DNA toxicity, disrupt lipid and protein glycosylation and inhibit telomerase. Therefore antiretroviral therapies target several pathways involved in accelerated or normal aging. Their combined effects are added to viral infection direct symptoms or to cell abnormalities induced by viral proteins.

Our multicentric (the 3 CISIH from Marseille, Nice and Montpellier) 3 year- long study will analyse 50 HIV1-infected naive patients (A group), apparied to 50 age- and sex-matched seronegative control subjects (recruited by CIC-UPCET of Marseille) and 100 HIV1-infected patients in first line of antiretroviral therapy for at least 12 months (B group). Patients of group A and B will be recruited in the 3 clinical unit. The HIV1- infected patients will be evaluated four times, at baseline, then every 12 months during 3 years. In case of initiation or changing of antiretroviral therapy, patients will be evaluated once more. Control subjects will be only evaluated at baseline.

Peripheral blood biological tests will be the following [Laboratory designation] : i/ viral load measurement, PBMC isolation, DNA extraction, proviral DNA measurement, cell and DNA storage [Virology, Timone CHU, Marseille]; ii/ assays of CD4, CD8, glycemia, insulinemia, HOMA, total-, LDL- and HDL-cholesterol, triglycerides [Biochemistry labs from the 3 CHU] ; iii/ antiretroviral drug assay (mass spectrometry) [Pharmacokinetics, Timone CHU, Marseille]; iv/ detection (western blotting, immunocytochemistry combined to image analysis of nuclear abnormalities) of PBMC nuclear, cytosolic and mitochondrial targets of antiretroviral drugs : A and B lamins, NF-B + I-B and proteasome activity assay, CD36 (glycosylation), mitochondrial Hsp70, ROS mitochondrial production, mitochondrial inner membrane potential, cytochrome C oxidase subunits 2 and 4 [Cell Biology, Timone CHU, Marseille] ; v/ genotyping the antiretroviral targets : lamin A (ZMPSTE24) and B (Rce1) processing proteases, Golgi SREBP-releasing proteases (MBTPS1 and S2), mitochondrial deoxynucleoside transporters (SLC25A4 to A6), mitochondrial proteases (MPPA, paraplegin) involved in processing of nuclear encoded proteins during their mitochondrial import ; quantitative PCR measurement of telomere length [Molecular Genetics, Timone CHU, Marseille]. Marseille's CIC-UPCET collaborated to the protocol design, will recruit control subjects and will be responsible for statistical treatment of data.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years and <65 years Able to give written consent Covered by French Social Security Non infected by HIV-2

* - A group HIV1-infected naive patients
* -B group infected patients in first line of antiretroviral therapy for at least 12 months
* -C group HIV seronegative Confirmed by a fast test of screening of the HIV at day one of study

Exclusion Criteria:

* Age < 18 years and > 65 years
* Not Able to give written consent
* Not Covered by French Social Security
* Infected by HIV-2
* treated by statin or biphosphonat amino
* concomitant treatment: diabetic or testosteron

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50 HIV1-infected naive patients (A group), apparied to 50 age- and sex-matched seronegative control (C group) subjects and 100 HIV1-infected patients in first line of antiretroviral therapy for at least 12 months (B group)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-04 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
lamin A measurement by western blotting

SECONDARY OUTCOMES:
Peripheral blood biological tests (cellular, molecular genetic)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle POIZOT-MARTIN, Principal Investigator — CHU Sainte Marguerite -Marseille; Marie-Pierre DROGOUL, Principal Investigator — CHU Sainte Marguerite -Marseille; Olivia FAUCHER, Principal Investigator — CHU Sainte Marguerite -Marseille; Amélie MENARD, Principal Investigator — CHU Sainte Marguerite -Marseille; Joëlle MICALLEF-ROLL, Principal Investigator — CHU Timone; Jacques REYNES, Principal Investigator — CISIH CHRU Gui de Chauliac- Montpellier; Pierre DELLAMONICA, Principal Investigator — CISIH CHU Nice; Pierre CAU, Principal Investigator — INSERM UMR S910 MARSEILLE; Catherine TAMALET, Principal Investigator — Laboratoire Virologie Marseille; Bruno LACARELLE, Principal Investigator — Unité INSERM U911 Marseille; Nicolas LEVY, Principal Investigator — Laboratoire Génétique Moléculaire Marseille; Patrick ROLL, Principal Investigator — Laboratoire biologie cellulaire Marseille
Locations (1):
- ANRS center from Marseille, Timone and Montpellier and Nice, Country of French, France

REFERENCES:
- [Derived] Perrin S, Cremer J, Faucher O, Reynes J, Dellamonica P, Micallef J, Solas C, Lacarelle B, Stretti C, Kaspi E, Robaglia-Schlupp A, Nicolino-Brunet C, Tamalet C, Levy N, Poizot-Martin I, Cau P, Roll P. HIV protease inhibitors do not cause the accumulation of prelamin A in PBMCs from patients receiving first line therapy: the ANRS EP45 "aging" study. PLoS One. 2012;7(12):e53035. doi: 10.1371/journal.pone.0053035. Epub 2012 Dec 28. PMID 23285253
- [Derived] Perrin S, Cremer J, Roll P, Faucher O, Menard A, Reynes J, Dellamonica P, Naqvi A, Micallef J, Jouve E, Tamalet C, Solas C, Pissier C, Arnoux I, Nicolino-Brunet C, Espinosa L, Levy N, Kaspi E, Robaglia-Schlupp A, Poizot-Martin I, Cau P. HIV-1 infection and first line ART induced differential responses in mitochondria from blood lymphocytes and monocytes: the ANRS EP45 "Aging" study. PLoS One. 2012;7(7):e41129. doi: 10.1371/journal.pone.0041129. Epub 2012 Jul 19. PMID 22829920
- See also: Related Info — http://anrs.fr